CLINICAL TRIAL: NCT07042347
Title: RCT of a Measurement Feedback App to Improve Data Quality, Supervision & Outcomes in Behavioral Health
Brief Title: Testing a Measurement Feedback App to Improve Data Quality, Supervision & Outcomes in Behavioral Health
Acronym: Footsteps
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 855228; R01MH136153 (NIH)
Record Dates: First submitted 2025-06-12; First posted 2025-06-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Autism; Challenging Behavior; ADHD; Oppositional Defiant Disorder
Keywords: data collection; Behavioral Health Technician (BHT); behavioral economics; implementation science; supervisory processes
MeSH Terms: conditions — Autistic Disorder; Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder

STUDY DESIGN:
Intervention Model Description: fully powered, randomized, hybrid type 2, pragmatic effectiveness-implementation mixed-methods trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Footsteps (Enhancements) (Experimental): An electronic platform for data collection ("Footsteps") that contains additional features designed to increase motivation to collect data and ease of data collection.
  Interventions: Behavioral: Behavioral economics strategies; Device: Electronic platform
- Data Collection Only App (No Enhancements) (Active Comparator): A basic electronic platform for data collection.
  Interventions: Device: Electronic platform

INTERVENTIONS:
Behavioral: Behavioral economics strategies — Behavioral economics features designed to increase motivation to collect data and ease of data collection on the electronic platform.
  Arms: Footsteps (Enhancements)
Device: Electronic platform — Electronic platform to collect data

SUMMARY:
The goal of this clinical trial is to test whether a smartphone-based data collection and feedback application ("Footsteps") improves the quality of behavioral data collected by one-to-one aides and leads to better youth mental health outcomes in school-aged youth (ages 4-17) who receive one-to-one support in schools.

The main questions it aims to answer are:

1. Does the Footsteps app improve aides' data collection quality (i.e., consistency, timeliness, and completeness)?
2. Does Footsteps use lead to improved youth behavioral health outcomes (e.g., SDQ, YTP, GAS scores)?
3. Does Footsteps improve communication and supervision processes between aides and clinical supervisors?

Researchers will compare aides using Footsteps to those using a "data collection only" control app to see if Footsteps leads to higher quality data collection, enhanced supervisory communication, and better youth outcomes.

Participants will:

* Use either Footsteps or a control app to record de-identified data on one client's behaviors and skills over 12 weeks
* Complete biweekly online surveys about data collection experiences, youth progress, and aide-supervisor communication
* Participate in a virtual intake and post-trial meeting
* (For a subset) Participate in a 30-45 minute qualitative interview about their experience using the app

ELIGIBILITY:
Inclusion Criteria:

* Aides must be employed by a community behavior health agency in Philadelphia or one of its surrounding counties
* and be working with at least one client in school who meets the following criteria: 1) between 4-17 years, 2) has a diagnosis associated with a challenging behavior (e.g., autism spectrum disorder, attention deficit hyperactivity disorder, oppositional defiant disorder) as indicated on their treatment plan, and 3) receiving 1:1 aide support.
* Supervisors must be employed by a community behavior health agency and supervise a participating aide. The investigators will recruit supervisors in dyads and not triads (i.e., no supervisors with two [or more] aides) to ensure there are 30 supervisor-aide dyads in total).

Exclusion Criteria:

* Aides who participated in the pilot trial of the Footsteps will be excluded from participating to recruit a sample naïve to Footsteps and the control app.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire total score | Assessed monthly (Baseline; Weeks 4, 8, and 12)
  A behavioral screening tool used to assess psychological attributes in children and adolescents, leading to a total score of 0 to 40. A higher total score indicates greater difficulties in emotional and behavioral functioning, while lower scores suggest fewer difficulties.
Data collection consistency | Assessed throughout 12-week trial
  an aggregate of the numbers of intervals scheduled, and the numbers of those intervals in which data was entered (% real time data)
Data collection timeliness | Assessed throughout 12-week trial
  for intervals in which data was entered, the time lag between occurrence and data entry

SECONDARY OUTCOMES:
Data collection completeness | Assessed throughout 12-week trial
  intervals classified as complete or incomplete according to whether the aide collected their planned metrics as required by their agency (% goals targeted)
Youth Top Problems | Assessed biweekly, at baseline through 12-week trial
  Top problems identified during intake meeting. Severity of each problem is rated from 0 (not a problem) to 4 (a very big problem). Severity ratings can be tracked for each problem individually or as an overall mean severity score created by averaging ratings from the same informant at the same measurement occasion
Goal Attainment Scaling | Assessed biweekly, at baseline through 12-week trial
  A method for measuring progress toward a goal, using a 5-point scale from -2 to +2. This scale helps quantify how well a goal was achieved, whether it was under-achieved, met, or over-achieved. Goals identified during intake meeting.

OTHER OUTCOMES:
Intentions for Implementors | Assessed biweekly, at baseline through 12-week trial
  The investigators adapted scales to measure mechanisms affecting data collection, including intentions, using social psychology methods (Armitage & Connor, 2001). The intentions measure had one item, which was rated from 1=strongly disagree to 7=strongly agree. Strongly agree meant stronger intentions to take data. Aides completed measures at baseline and post-trial (3 weeks). Data reported are changes over time.
Attitudes for Implementors | Assessed biweekly, at baseline and through 12-week trial
  The investigators adapted scales to measure mechanisms affecting data collection, including attitudes, using social psychology methods (Armitage & Connor, 2001). The attitudes measure had one item, which was rated from 1=good to 7=bad (meaning that taking data would be bad). Attitudes had 2 items. These items were averaged to create the scale score which could range from 1 to 7 for each measure. Aides completed measures at baseline and post-trial (3 weeks). Data reported are changes over time.
Perceived Norms for Implementors | Assessed biweekly, at baseline through 12-week trial
  The investigators adapted scales to measure mechanisms affecting data collection, including perceived norms, using social psychology methods (Armitage & Connor, 2001). The perceived norms measure had one item, which was rated from 1=strongly disagree to 7=strongly agree. Strongly agree meant stronger influence of norms on taking data. Aides completed measures at baseline and post-trial (3 weeks). Data reported are changes over time.
Descriptive Norms for Implementors | Assessed biweekly, at baseline through 12-week trial
  The investigators adapted scales to measure mechanisms affecting data collection, including descriptive norms, using social psychology methods (Armitage & Connor, 2001). The perceived norms measure had one item, which was rated from 1=strongly disagree to 7=strongly agree. Strongly agree meant stronger influence of norms on taking data. Aides completed measures at baseline and post-trial (3 weeks). Data reported are changes over time.
Self-Efficacy for Implementors | Assessed biweekly, at baseline through 12-week trial
  The investigators adapted scales to measure mechanisms affecting data collection, including self-efficacy, using social psychology methods (Armitage & Connor, 2001). The self-efficacy measure had one item, which was rated from 1=strongly disagree to 7=strongly agree. Strongly agree meant stronger self-efficacy about taking data. Self-Efficacy had 2 items. These items were averaged to create the scale score which could range from 1 to 7 for each measure. Aides completed measures at baseline and post-trial (3 weeks). Data reported are changes over time.
System Usability Scale | Assessed at post-trial (Week 12)
  The investigators used the System Usability Scale (SUS; Brooke, 1996) to measure aides' reactions to various statements regarding the app's usability with 10 items that use a 5-point scale from (1) strongly disagree to (5) strongly agree. The SUS has high internal consistent reliability (Cronbach's alpha = .91) and demonstrated sensitivity to change (Lewis, 2018). The investigators adapted the original questionnaire to replace "system" with "app" across all items. The SUS is calculated as a proportion score out of 100, with higher scores indicating higher usability (≥85 = Excellent; ≥71 = Good; ≥51 = Okay (Bangor et al.).
Supervisor <> Aide Communication | Assessed biweekly, at baseline through 12-week trial
  The investigators will compare the groups on combined frequency and content of the communications by using a three-level ordinal response for each period (0=no communication, 1=communication, with discussion of client, 2=communication, discussion of client, and discussion of treatment strategy changes).

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Nuske, PhD, Principal Investigator — University of Pennsylvania; David Mandell, Sc.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nuske HJ, Buck J, Ramesh B, Becker-Haimes EM, Zentgraf K, Mandell DS. Making Progress Monitoring Easier and More Motivating: Developing a Client Data Collection App Incorporating User-Centered Design and Behavioral Economics Insights. Soc Sci (Basel). 2022 Mar;11(3):106. doi: 10.3390/socsci11030106. Epub 2022 Mar 3. PMID 35496358
- See also: Website which describes the development of this application and available features. — https://www.digitalmentalhealth.org/footsteps